CLINICAL TRIAL: NCT05621941
Title: A Strategy Game Supporting Goal Management Training Intervention for the Treatment of Executive Problems After Acquired Brain Injury: a Randomized Controlled Pilot Study for Usability and Preliminary Efficacy
Brief Title: Strategy Game Supporting Goal Management Training Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klimmendaal Revalidatiespecialisten (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Karman Line GMT; Dutch Trial Register (Registry Identifier: NL9200)
Record Dates: First submitted 2022-11-04; First posted 2022-11-18 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Acquired Brain Injury; Executive Dysfunction; Neuropsychological Rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game-Supported Goal Management Training (Experimental): Seven treatment sessions given once a week (60 minutes) under guidance of a clinical neuropsychologist and cognitive trainer or occupational therapist.
  Interventions: Behavioral: Game-Supported Goal Management Training
- Information Group (Active Comparator): Seven information sessions given once a week (60 minutes) under guidance of a clinical neuropsychologist.
  Interventions: Behavioral: Information Group

INTERVENTIONS:
Behavioral: Game-Supported Goal Management Training — The investigational treatment is based on a compensatory strategy training named Goal Management Training (GMT). The investigational treatment will include GMT in combination with a compensatory strategy game which allows the patient to learn and apply the algorithm of GMT in a safe and controlled environment. This means that the multiple steps of the GMT will be learned during the treatment sessions under guidance of a therapist as well as in their own home environment by using the compensatory strategy game.
  Arms: Game-Supported Goal Management Training
Behavioral: Information Group — In the information group, patients are informed about non-specific consequences of acquired brain injury, aimed to increase patient's insight into their condition and with that improving functioning. The program consists of the following subjects: 1) cause of brain injury, 2) information processing and attention, 3) memory, 4) planning and performance, 5) fatigue, 6) changes in emotion and behavior and 7) processing and adjustments.
  Arms: Information Group

SUMMARY:
Many brain-injured patients referred for outpatient rehabilitation have difficulties with planning, problems solving, and reasoning. These difficulties can be characterized as executive deficits, which can vary from relatively mild to rather severe. Executive deficits lead to real-life everyday disorganization and difficulties in instrumental activities of daily living (IADL tasks). Goal Management Training (GMT) is a successful treatment for executive deficits and helps to structure activities in daily life. GMT entails learning and applying an algorithm, in which a daily task is subdivided into multiple steps to handle executive difficulties of planning, and problem solving. Patients are taught compensatory strategies not to strengthen the executive functions, but to enable them to minimize disabilities and participation problems and to function more independently in daily life. The currently implemented GMT treatment in the Netherlands is aimed at relearning two specific tasks. However, to adopt the GMT strategy and ensure maximal profitability for patients, they have to learn to use the algorithm in different situations and tasks, which requires a comprehensive, time-consuming and thus labour-intensive treatment. Along with this, brain games become increasingly attractive as an (add-on) intervention, most notably in an effort to develop home-based personalized care, and because of their machine learning algorithms which tailors the game to the level of the individual player. Until now, however, the rationale behind brain games is based on what can be considered the restorative approach (i.e. strengthening of executive problems) rather than practicing compensatory strategies, with no transfer to improvements in daily life functioning. The present study fills a gap in the literature by investigating a new developed treatment that incorporates GMT and a treatment supporting strategy game in a pilot sample of brain injured patients. The primary objective of this pilot study is to obtain an efficacy estimate and investigate the feasibility of GMT with a new game that incorporates strategy training in improving executive functions in a pilot sample of brain-injured patients. This study investigates usability and acceptability of our new developed GMT treatment to brain-injured patients in the chronic phase (>3 months post-onset), and obtains an efficacy estimate, focusing on transfer of treatment effects to untrained (instrumental) activities of daily living. Chronic brain-injured patients will be allocated to the game-supported GMT treatment or to an information group using block randomization. It will be an assessor blind study in which researchers responsible for assessing or analyzing data will be blind for the received treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any type of acquired brain injury of non-progressive nature in the past, being more than three months post injury.
* A Clinically meaningful score of executive complaints on the BRIEF-A.
* Aged between 18 and 70 years
* Referred for outpatient rehabilitation
* Living independently at home

Exclusion Criteria:

* Inability to speak/ understand the Dutch language
* Co-morbidity that might affect outcome (e.g. neurodegenerative disorders, aphasia, neglect, and major psychiatric illness)
* Substance abuse
* No access to a smartphone, laptop or tablet
* Unable to look at a computer screen for 15 minutes
* Being unable to operate a keyboard or computer mouse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance on untrained IADL tasks immediately after the intervention | Baseline and immediately after the intervention
  Standardized scale measuring performance of an untrained IADL task (int. al. the percent change in the number of correct steps) before (baseline) and after treatment (post treatment). The untrained IADL tasks will be divided into multiple steps using the GMT method. These steps will be assessed using four categories: 1) additional/unrelated; 2) absent/incomplete; 3) questionable/ineffective; 4) competent/correct, using task-specific assessment forms.

SECONDARY OUTCOMES:
Change from baseline Goal Attainment Scaling (GAS) on untrained task performance immediately after the intervention | Baseline and immediately after the intervention
  Quantifying the subjective improvement on untrained task performance
Change from baseline subjective strategy use immediately after the intervention | Baseline and immediately after the intervention
  The subjective experience of strategy use in daily life and during the performance of IADL tasks, as measured by two short self-reported questionnaires.
Change from baseline participation as measured by the USER-P immediately after the intervention | Baseline and immediately after the intervention
  "Utrecht Scale for Evaluation of Rehabilitation - Participation" (USER-P)
Change from baseline executive functioning as measured with the Zoo map test immediately after the intervention | Baseline and immediately after the intervention
  Zoo map test
Change from baseline executive functioning as measured with the modified six elements test immediately after the intervention | Baseline and immediately after the intervention
  Modified six elements test
Change from baseline executive functioning as measured with the Brixton immediately after the intervention | Baseline and immediately after the intervention
  Brixton
Change from baseline subjective cognitive complaints as measured with the Cognitive Failure Questionnaire (CFQ) immediately after the intervention | Baseline and immediately after the intervention
  Cognitive Failure Questionnaire (CFQ)
Change from baseline executive functioning as measured with the OxMET-NL immediately after the intervention | Baseline and immediately after the intervention
  Oxford Multiple Errands Test - Dutch version (OxMET-NL)
Change from baseline subjective executive complaints immediately after the intervention | Baseline and immediately after the intervention
  Behavior Rating Inventory of Executive Function- Adult Version (BRIEF-A)
Change from baseline Goal Attainment Scaling (GAS) on treatment goals immediately after the intervention | Baseline and immediately after the intervention
  Quantifying the achievement of treatment goals, only measured in the game-supported GMT group.
System Usability Scale (SUS) questionnaire | Immediately after the intervention
  To evaluate the usability of the game-supported GMT treatment.
Technological Acceptance Model (TAM) questionnaire | Immediately after the intervention
  To evaluate the user-acceptance of the game-supported GMT treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Klimmendaal Revalidatiespecialisten, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://trialsearch.who.int/Trial2.aspx?TrialID=NL9200